CLINICAL TRIAL: NCT05716438
Title: Prospective Evaluation of Loss of Reduction and Cast Parameters Following Cast Bivalving for Pediatric Distal Radius Fractures
Brief Title: Prospective Evaluation of Cast Bivalving for Pediatric Distal Radius Fractures
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Daniel Cognetti, Primary Investigator, Brooke Army Medical Center
Other Study IDs: 2019.008
Record Dates: First submitted 2023-01-15; First posted 2023-02-08 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-01

CONDITIONS: Distal Radius Fracture; Loss of Anatomical Alignment After Fracture Reduction
Keywords: Cast; Pediatric; Cast Index; Distal Radius Fracture; Loss of Reduction; Bivalve
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Forearm anteroposterior and lateral plain radiograph — 2 view plain film of forearm after valving a short arm cast.

SUMMARY:
Pediatric patients with distal radius fractures are most commonly treated non-operatively with fracture reduction and cast immobilization. In order to prevent complications from increased swelling after the injury (or fracture manipulation) casts may be split along their length to relieve pressure. However, this can compromise the casts' structural integrity, predisposing fractures to loss of reduction. The goal of this study was to investigate if cast bivalving, or splitting the cast longitudinally on both sides, resulted in any immediate change to bony alignment and to assess if bivalving effected cast parameters associated with loss of reduction.

DETAILED DESCRIPTION:
Displaced pediatric distal radius fractures are treated with fracture reduction and cast immobilization. Currently, at our institution (and many others) radiographic assessment to determine acceptable fracture alignment and cast parameters is done immediately after cast application. However, afterward casts are often split on both sides along their length, in a process known as bivalving, prophylactically treating for post-traumatic soft tissue edema. While bivalving is felt to relieve pressure from the cast, it may also diminish the structural integrity of the cast. Although it is well-established that loss of fracture alignment is most common in the first few weeks after fracture reduction there have been no studies to evaluate any immediate changes to fracture reduction or cast parameters that may occur after bivalving. Thus, the goal of this study was to assess if pediatric distal radius fracture alignment was affected by cast bivalving by obtaining post-bivalve radiographs in addition to standard post-cast radiographs.

ELIGIBILITY:
Inclusion Criteria:

* Guardian must be present
* Able/eligible to complete follow-up
* Initial injury within 72 hours
* Distal Radius fracture with or without distal ulna fracture
* Requiring non-operative management with molded cast

Exclusion Criteria:

* Open fractures
* Re-fractures
* Pathologic fractures
* Fractures associated with neurovascular injury
* Poly trauma incident
* Intubated patients or unable to verbalize symptoms of pain
* Preexisting medical history that effects musculoskeletal health

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Pediatric patients with displaced distal radius fractures requiring reduction presenting to Brooke Army Medical Center within 72 hours of injury.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2023-04-20 (Estimated)

PRIMARY OUTCOMES:
Change in reduction after bivalving | up to 24 hours
  Change in fracture reduction of 2mm or 5 degrees in angulation on radiographs after bivalving
Change in reduction at follow-up | up to 30 days
  Change in fracture reduction of 2mm or 5 degrees in angulation on radiographs at follow-up
Cast Index | through study completion, up to 2 years
  Cast index, the ratio of sagittal to coronal width from the inside edges of the cast at the fracture site will be measured via radiographs.
Gap Index | through study completion, up to 2 years
  Gap index is a measure of space between the cast and skin measured as a ratio to the inside diameter of the cast, assessed at the level of the fracture on anteroposterior and lateral radiographs.
Three Point Index | through study completion, up to 2 years
  Three point index, a measure of space between the cast and skin at sites of the three point mold, with reference to the adequacy of reduction, assessed via the contact length of the proximal and distal fracture segments on anteroposterior and lateral radiographs.

OTHER OUTCOMES:
Complications | through study completion, up to 2 years
  Surgical intervention, cast saw burns, physeal arrest, refracture (after enrollment)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Cognetti, MD, Principal Investigator — Brooke Army Medical Center
Locations (1):
- Brooke Army Medical Center, Fort Sam Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided